CLINICAL TRIAL: NCT05318105
Title: A Randomized Controlled Study to Evaluate the Safety and Effectiveness of the Aquadex System in Patients With Heart Failure and Fluid Overload
Brief Title: Ultrafiltration Versus IV Diuretics in Worsening Heart Failure
Acronym: REVERSE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN07687
Record Dates: First submitted 2022-03-10; First posted 2022-04-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure (for Example, Fluid Overload); Heart Failure; Fluid Overload
Keywords: Heart failure; Fluid overload
MeSH Terms: conditions — Heart Failure; Edema | interventions — Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aquadex ultrafiltration therapy (Experimental)
  Interventions: Device: Aquadex Smartflow® System
- IV loop diuretics (Active Comparator)
  Interventions: Drug: IV Loop Diuretics

INTERVENTIONS:
Device: Aquadex Smartflow® System — ultrafiltration
  Arms: Aquadex ultrafiltration therapy
Drug: IV Loop Diuretics — diuretics
  Arms: IV loop diuretics

SUMMARY:
The REVERSE-HF study is a randomized controlled trial to evaluate clinical outcomes of adjustable ultrafiltration with the Aquadex System as compared to adjustable IV loop diuretics in patients with worsening heart failure (HF) and fluid overload.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Man, or non-pregnant woman
* Admitted to the hospital with a diagnosis of acute decompensated heart failure
* On regularly prescribed oral loop diuretics, Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors or a Mineralcorticoid Receptor Antagonists (MRA) prior to admission
* Fluid overload manifested by at least three clinical indications (e.g., edema, an excess of at least 10 pounds of fluid, etc.)
* Provide written informed consent

Exclusion Criteria:

* New diagnosis of heart failure
* Acute coronary syndromes
* Creatinine ≥ 3.0 mg/dl or planned renal replacement therapies at the time of enrollment
* Contraindications to systemic anticoagulation
* Severe concomitant disease expected to prolong hospitalization or cause death in less than 90 days
* Sepsis or ongoing systemic infection
* Active myocarditis
* Constrictive pericarditis or restrictive cardiomyopathy
* Severe aortic stenosis
* Any condition in the opinion of the investigator that would prevent the patient from follow-up/survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first heart failure (HF) event | within 30 days
  Heart Failure (HF) event defined as any HF rehospitalization or unplanned use of IV loop diuretics, vasoactive medications or Aquadex therapy in any outpatient setting.

SECONDARY OUTCOMES:
Win ratio analysis | within 30 days
  Win ratio analysis of cardiovascular (CV) mortality, HF events and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sean Pinney, MD, Principal Investigator — Mount Sinai Morningside; Maria DeVita, MD, FASN, Principal Investigator — Lenox Hill Hospital
Locations (17):
- United States (17):
  - Banner Health, Tucson, Arizona
  - MemorialCare, Long Beach Medical Center, Long Beach, California
  - Sharp Memorial Hospital, San Diego Cardiac Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - BayCare Medical Group, Morton Plant, Clearwater, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Health, Detroit, Michigan
  - Mount Sinai Morningside, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Northwell Health, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Abington Jefferson Health, Abington, Pennsylvania
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Sentara Norfolk General Heart Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCallum W, Sarnak MJ. Cardiorenal Syndrome in the Hospital. Clin J Am Soc Nephrol. 2023 Jul 1;18(7):933-945. doi: 10.2215/CJN.0000000000000064. Epub 2023 Jan 13. PMID 36787124